CLINICAL TRIAL: NCT01277900
Title: Efficacy and Safety Study of LRYGB to Treat Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) to Treat Type 2 Diabetes Mellitus
Acronym: ADSMT-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asia Metabolic Surgery Research Group (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Dr. Huang, Chih-Kun, Bariatric & Metabolic International Surgery Center
Other Study IDs: ADSMT-1
Record Dates: First submitted 2011-01-11; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus - Poor Control

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laparoscopic Roux-en-Y gastric bypass: Laparoscopic Roux-en-Y gastric bypass will be used as a standard procedure to treat type 2 diabetes mellitus
  Interventions: Procedure: Laparoscopic Roux en Y gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Roux en Y gastric Bypass — Laparoscopic Roux-en-Y gastric bypass will be used as a standard procedure to treat type 2 diabetes mellitus
  Other Names: LRYGB

SUMMARY:
Type 2 diabetes mellitus (T2DM) resolution in morbidly obese patients following bariatric surgery suggests the efficacy of metabolic surgery in non-morbidly obese patients (body mass index [BMI]<35 kg/m2). Many researches have shown available evidence about the efficacy and safety of metabolic surgery for resolution of T2DM in the non-morbidly obese. One of the most effective metabolic surgeries is laparoscopic Roux-en-Y gastric bypass (LRYGB). The investigators intend to run a 3 year prospective multicenter study to evaluate the remission efficacy of laparoscopic Roux-en-Y gastric bypass in Type 2 Diabetes mellitus with low BMI (BMI:25-35) in Asia area.

DETAILED DESCRIPTION:
The study is designed including 9 bariatric centers across Asia region( China, Korea, Phillipine, Singapore and Taiwan). Totally 500 patients with confirmed diagnosis of T2DM and BMI between 25-35 kg/m2 will be enrolled from January 2011 to December 2013. Preoperative surgical parameters, blood, biochemistry data, gastrointestinal hormones, upper gastrointestinal studies, abdominal ultrasound, peri-operative & postoperative complications will all be recorded and analyzed. Patient inclusion criteria: 1.) T2DM diagnosed over 1 year; 2.) age ranged 30-60 years; 3.) BMI 25-35 kg/m2; 4.) Patient consent and will to receive long-term follow up and periodic check up. Exclusion criteria: 1.) T1DM; 2.) Substance abuse; 3.) Planned pregnancy within 2 year after surgery; 3.) Uncontrolled psychiatric disease; 4.) Lost follow up. Institutions inclusion criteria: Professional experience over 30 LRYGB performed. Trial termination criteria: Surgical mortality over 0.5% in the first year, and Diabetes remission rate failure over 20% in one year.

All data will be collected yearly in one center. The analysis of parameter, statistics and brief results will be informed to enrolled institutions periodically.

ELIGIBILITY:
Inclusion Criteria:

1. T2DM diagnosed over 1 year;
2. Age ranged 30-60 years;
3. BMI 25-35 kg/m2;
4. Patient consent and will to receive long-term follow up and periodic check up.

Exclusion Criteria:

1. T1DM;
2. Substance abuse;
3. Planned pregnancy within 2 year after surgery;
4. Uncontrolled psychiatric disease;
5. Lost follow up.

Institutions inclusion criteria: Professional experience over 30 LRYGB performed.

Trial termination criteria: Surgical mortality over 0.5% in the first year, and Diabetes remission rate failure over 20% in one year.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 500 type 2 diabetes mellitus patients with BMI between 25-35 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Gastric Bypass in the Treatment of Type 2 Diabetes in Patients with a BMI of 25 to 35 kg/m2 | 3 years (from 2011 to 2013)
  An observational, prospective and multi-center study will be carry out with IRB approval. A total of 500 type 2 diabetes mellitus patients with low BMI (25-35 kg/m2) will be collected in different surgical institutions. Pre and post operative biochemical parameters will be collected at the 1st, 6th, 12th, 24th and 36th months. Comparative outcomes will support the relationship between diabetes improvement or remission and the surgical intervention.
  Blood parameters: CBC, hs-CRP, SMA12, HbA1c, Fasting C-peptide, Insulin, OGTT,C-peptide and DM antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Kun Huang, Doctor, Principal Investigator — E-DA Hospital
Locations (1):
- BMI Surgery Center, E-DA Hospital, Kaohsiung, Taiwan, Taiwan